CLINICAL TRIAL: NCT03348150
Title: Treatment of Peritoneal Dissemination in Stomach Cancer Patients With Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy (HIPEC).
Brief Title: Gastrectomy + Cytoreductive Surgery + HIPEC for Gastric Cancer With Peritoneal Dissemination.
Acronym: PERISCOPEII
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Erasmus Medical Center (Other); UMC Utrecht (Other); University Medical Center Groningen (Other); Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M15PEC; 2015-005695-15 (EudraCT Number); NL56123.031.15 (Other: CCMO)
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Stomach Neoplasm; Peritoneal Carcinomatosis
Keywords: HIPEC; Hyperthermic Intraperitoneal Chemotherapy; gastrectomy; cytoreductive surgery; oxaliplatin; docetaxel
MeSH Terms: conditions — Stomach Neoplasms; Peritoneal Neoplasms | interventions — Cytoreduction Surgical Procedures; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gastrecomy + Cytoreductive surgery + HIPEC (Experimental): Gastrectomy combined with cytoreductive surgery and HIPEC (experimental treatment)
  Interventions: Procedure: Cytoreductive surgery + Gastrecomy; Drug: Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
- palliative systemic chemotherapy (No Intervention): Palliative systemic chemotherapy only (standard treatment)

INTERVENTIONS:
Procedure: Cytoreductive surgery + Gastrecomy — Complete cytoreduction followed by a (sub)total gastric resection with D2 lymphadenectomy.
  Arms: Gastrecomy + Cytoreductive surgery + HIPEC
Drug: Hyperthermic Intraperitoneal Chemotherapy (HIPEC) — HIPEC: perfusion with oxaliplatin (460mg/m2 ) (42 °C) followed by docetaxel (50mg/m2 ) (37°C)
  Other Names: HIPEC
  Arms: Gastrecomy + Cytoreductive surgery + HIPEC

SUMMARY:
A randomized controlled two-armed phase III trial for gastric cancer patients with peritoneal dissemination. Randomization between gastrectomy + cytoreductive surgery + HIPEC (experimental arm) and palliative systemic chemotherapy (standard arm).

DETAILED DESCRIPTION:
Rationale: For gastric cancer patients with peritoneal carcinomatosis palliative systemic chemotherapy is the standard treatment in the Netherlands. There are no potentially curative treatment options. Peritoneal carcinomatosis, in contrast to lymphatic and haematogenous dissemination, should be regarded as locoregional extension of disease. Administering chemotherapeutic drugs directly into the peritoneal cavity has an advantage over systemic chemotherapy since high concentrations of cytotoxic drugs can be delivered directly into the peritoneal cavity with little systemic toxicity. The combination of intraperitoneally administered chemotherapy with cytoreductive surgery and a radical gastrectomy has shown promising results in gastric cancer patients in Asia. As with other gastric cancer issues, the results obtained in Asian patients cannot be extrapolated directly to Western patients.

Objective: The primary aim of this study is to compare the overall survival between gastric cancer patients with limited peritoneal carcinomatosis and/ or tumour positive peritoneal cytology treated with gastrectomy, cytoreductive surgery and HIPEC and those treated with the current standard treatment, i.e. palliative systemic chemotherapy.

Study design : This is a multicentre randomised controlled two-armed phase III trial. Patients will be randomised (1:1) between palliative systemic chemotherapy only (standard treatment) and gastrectomy combined with cytoreductive surgery and HIPEC (experimental treatment).

Study population: Gastric cancer patients are eligible for inclusion if (1) the primary cT3-cT4 gastric tumour including regional lymph nodes is considered to be resectable, (2) limited peritoneal carcinomatosis (<7) and/ or tumour positive cytology is confirmed by laparoscopy or laparotomy, and (3) systemic chemotherapy (prior to inclusion) was without disease progression.

Main study parameters/endpoints: The study sample size (182 patients) is calculated from the hypothesis that the median overall survival of the patients treated according to protocol in the experimental arm is 18 months, as compared to a median overall survival of 10 months in the standard arm. Statistical analysis will be done according to the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Biopsy proven primary adenocarcinoma (or undifferentiated carcinoma) of the stomach. Including tumours at the oesophagogastric junction provided that the bulk of the tumour is located in the stomach, and, the intended surgical treatment is a gastric resection and not an oesophagectomy. A high intra-thoracic anastomosis is allowed, but not if a thoracotomy is necessary.
* cT3-cT4 tumour (TNM classification, 7th edition), considered to be resectable (including lymph nodes)
* Limited peritoneal carcinomatosis (PCI <7) and/ or tumour positive peritoneal cytology confirmed by laparoscopy or laparotomy and proven by pathological examination
* Treatment with systemic chemotherapy, with the latest course ending within 8 weeks prior to inclusion. All currently standard chemotherapy regimens are acceptable
* Absence of disease progression during systemic chemotherapy (prior to inclusion)
* WHO performance status 0-2
* Adequate bone marrow, hepatic and renal function. Minimally acceptable laboratory values at start of the study inclusion:

  * ANC ≥ 1.5 x 109 /L
  * Platelet count ≥ 100 x 109 /L
  * Serum bilirubin ≤ 1.5 x ULN, and ALAT and ASAT ≤ 2.5 x ULN
  * Creatinine clearance ≥ 50 ml/min (measured or calculated by Cockcroft-Gault formula)
* For female patients who are not sterilised or in menopause (i.e., amenorrhea ≥1 year if age ≥60 years, or ≥2 years if age <60 years):

  * negative pregnancy test (urine/serum)
  * no breast feeding or active pregnancy ambition
  * reliable contraceptive methods
* Signed informed consent

Exclusion Criteria:

* Distant metastases (e.g., liver, lung, para-aortic lymph nodes; i.e., stations 14 and 16) or small bowel dissemination
* Recurrent gastric cancer
* Prior resection of the primary gastric tumour
* Non-synchronous peritoneal carcinomatosis
* Current other malignancy (other than cervix carcinoma and basalioma)
* Uncontrolled infectious disease or known infection with Human Immunodeficiency Virus type -1 or -2
* A known history of hepatitis B or C with active viral replication
* Recent myocardial infarction (< 6 months) or unstable angina
* Any medical condition not yet specified above that is considered to interfere with study procedures, including adequate follow-up and compliance and/or would jeopardise safe treatment
* Known hypersensitivity for any of the applied chemotherapeutic agents and/or their solvents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2025-09-17 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years
  To compare the overall survival between gastric cancer patients with limited peritoneal carcinomatosis and/ or tumour positive peritoneal cytology treated with gastrectomy, cytoreductive surgery and HIPEC and those treated with the current standard treatment, i.e. palliative systemic chemotherapy.

SECONDARY OUTCOMES:
progression free survival | 5 years
  To compare the progression free survival between gastric cancer patients with limited peritoneal carcinomatosis and/ or tumour positive peritoneal cytology treated with gastrectomy, cytoreductive surgery and HIPEC and those treated with the current standard treatment, i.e. palliative systemic chemotherapy.
treatment-related toxicity | 5 years
  To study treatment-related toxicity in gastric cancer patients with limited peritoneal carcinomatosis and/ or tumour positive peritoneal cytology treated with gastrectomy, cytoreductive surgery and HIPEC.
costs and health benefits | 5 years
  To compare the costs and health benefits of a gastrectomy in combination with cytoreductive surgery and HIPEC, to the costs and health benefits of standard palliative systemic chemotherapy in patients with limited peritoneal carcinomatosis and/ or tumour positive peritoneal cytology.

CONTACTS AND LOCATIONS:
Overall Officials: Johanna van Sandick, MD, PHD, Principal Investigator — Surgeon
Locations (1):
- Antoni van Leeuwenhoek/ Netherlands Cancer institute, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Kaaij RT, Braam HJ, Boot H, Los M, Cats A, Grootscholten C, Schellens JH, Aalbers AG, Huitema AD, Knibbe CA, Boerma D, Wiezer MJ, van Ramshorst B, van Sandick JW. Treatment of Peritoneal Dissemination in Stomach Cancer Patients With Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy (HIPEC): Rationale and Design of the PERISCOPE Study. JMIR Res Protoc. 2017 Jul 13;6(7):e136. doi: 10.2196/resprot.7790. PMID 28705789
- [Derived] Koemans WJ, van der Kaaij RT, Boot H, Buffart T, Veenhof AAFA, Hartemink KJ, Grootscholten C, Snaebjornsson P, Retel VP, van Tinteren H, Vanhoutvin S, van der Noort V, Houwink A, Hahn C, Huitema ADR, Lahaye M, Los M, van den Barselaar P, Imhof O, Aalbers A, van Dam GM, van Etten B, Wijnhoven BPL, Luyer MDP, Boerma D, van Sandick JW. Cytoreductive surgery and hyperthermic intraperitoneal chemotherapy versus palliative systemic chemotherapy in stomach cancer patients with peritoneal dissemination, the study protocol of a multicentre randomised controlled trial (PERISCOPE II). BMC Cancer. 2019 May 6;19(1):420. doi: 10.1186/s12885-019-5640-2. PMID 31060544